CLINICAL TRIAL: NCT07330999
Title: Comparison of Standard PENG Block Versus PENG With Perineural Dexamethasone or Perineural Dexmedetomidine in Patients Aged 65 Years and Older Undergoing Hip Surgery: A Randomized Controlled Trial
Brief Title: Three Variants of the PENG Block With and Without Perineural Adjuvants in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medications will be prepared by a clinician not involved in patient care or outcome assessment. All participants will receive identical appearing syringes and identical volumes of perineural and intravenous solutions containing either active medication or normal saline placebo. Patients, care providers, investigators, and outcome assessors will remain blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block With Ropivacaine Only (Control) (Active Comparator): Participants will receive a Pericapsular Nerve Group (PENG) block using 20 mL of 0.2% ropivacaine without any adjuvant administered perineurally or intravenously. All participants will receive standard perioperative care and multimodal analgesia. Ondansetron will be used as standard prophylaxis for postoperative nausea and vomiting.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- PENG Block With Perineural Dexamethasone (Active Comparator): Participants will receive a PENG block using 20 mL of 0.2% ropivacaine combined with 4 mg of dexamethasone administered perineurally. No dexamethasone will be given intravenously. All participants will receive standard perioperative care and multimodal analgesia.
  Interventions: Drug: Dexamethasone 4mg
- PENG Block With Perineural Dexmedetomidine (Active Comparator): Participants will receive a PENG block using 20 mL of 0.2% ropivacaine combined with 25 µg of dexmedetomidine administered perineurally. No dexamethasone will be given intravenously. All participants will receive standard perioperative care and multimodal analgesia.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — 20 mL of 0.2% ropivacaine administered perineurally as part of the PENG block. No perineural or intravenous adjuvant drugs will be used in this arm.
  Arms: PENG Block With Ropivacaine Only (Control)
Drug: Dexamethasone 4mg — 4 mg of dexamethasone administered perineurally together with 20 mL of 0.2% ropivacaine for the PENG block. No intravenous dexamethasone will be administered.
  Arms: PENG Block With Perineural Dexamethasone
Drug: Dexmedetomidine — 25 micrograms of dexmedetomidine administered perineurally together with 20 mL of 0.2% ropivacaine for the PENG block. No intravenous dexamethasone will be administered.
  Arms: PENG Block With Perineural Dexmedetomidine

SUMMARY:
This study will compare three versions of the Pericapsular Nerve Group (PENG) block in adults aged 65 years and older who are undergoing hip surgery. The PENG block is a regional anesthesia technique used to reduce pain around the hip joint and may improve early recovery after surgery.

All patients in the study will receive the PENG block using 20 mL of 0.2% ropivacaine. They will then be randomly assigned to one of three groups:

Group 1: PENG block using ropivacaine only (no additional medications). Group 2: PENG block using ropivacaine with 4 mg of dexamethasone injected near the nerves.

Group 3: PENG block using ropivacaine with 25 micrograms of dexmedetomidine injected near the nerves.

Dexamethasone and dexmedetomidine are medications that may increase the duration and quality of regional anesthesia. It is not known whether adding one of these medications provides longer-lasting or better pain relief compared to using ropivacaine alone.

The main purpose of this study is to determine whether the addition of dexamethasone or dexmedetomidine improves the effectiveness of the PENG block in relieving pain after hip surgery. The study will evaluate pain levels, opioid consumption, time to first rescue pain medication, need for additional analgesia, and recovery outcomes. Safety, side effects, and any block-related complications will also be monitored.

We hypothesize that adding either perineural dexamethasone or dexmedetomidine will result in longer and more effective pain relief compared with the standard PENG block without an adjuvant.

This research may help identify the most effective form of the PENG block for older adults undergoing hip surgery and contribute to improved pain management, reduced opioid use, and better postoperative recovery.

DETAILED DESCRIPTION:
Hip surgery in older adults is frequently associated with significant postoperative pain, delayed mobilization, and increased opioid requirements. Poor pain control in this population can lead to complications such as delirium, prolonged hospitalization, reduced physical function, and slower rehabilitation. Effective regional anesthesia may improve safety and recovery after hip surgery.

The Pericapsular Nerve Group (PENG) block is a relatively new regional anesthesia technique designed to target the sensory innervation of the hip joint while preserving motor function. This motor-sparing feature may allow earlier mobilization and reduce the negative effects of immobilization in older patients.

Ropivacaine is the standard local anesthetic commonly used in peripheral nerve blocks. Small doses of adjuvant medications such as dexamethasone or dexmedetomidine may prolong the duration of analgesia and improve the quality of pain control. However, it remains unclear whether the addition of these medications provides any clinically meaningful benefit when used with the PENG block in older adults. There is also limited evidence directly comparing different adjuvants to a standard PENG block without additional medication.

This randomized controlled trial will compare three variants of the PENG block in adults aged 65 years and older undergoing hip surgery. All participants will receive a PENG block with 20 mL of 0.2% ropivacaine. They will then be randomly assigned to one of three groups:

Standard PENG block with ropivacaine alone (no adjuvant). PENG block with 4 mg of perineural dexamethasone. PENG block with 25 micrograms of perineural dexmedetomidine. All patients will receive standard perioperative care and multimodal analgesia. The study will assess pain scores, time to first rescue analgesia, total opioid consumption, functional mobility, incidence of postoperative nausea and vomiting, block duration, motor function, and complications. Safety will also be monitored, including block-related and neurological adverse events.

The primary objective of this study is to determine whether perineural dexamethasone or dexmedetomidine improves postoperative analgesia compared with a standard PENG block without adjuvant. We hypothesize that both adjuvants may prolong analgesia and reduce opioid requirements, but their effectiveness and safety profile may differ.

This study aims to provide evidence that can help guide anesthesiologists in selecting the optimal variant of the PENG block for older adults undergoing hip surgery, intending to improve postoperative pain control, support early rehabilitation, and reducing complications associated with opioid use and delayed mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective or emergency hip surgery (e.g., hip fracture fixation or hip arthroplasty)
* ASA physical status I-III
* Planned use of a PENG block as part of perioperative analgesia
* Ability to communicate pain intensity using the NRS scale
* Written informed consent obtained from the patient or legal representative

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Known allergy, intolerance, or contraindication to any of the study medications: ropivacaine, dexamethasone, dexmedetomidine
* Pre-existing neurological deficit or neuropathy in the affected limb
* Coagulopathy or laboratory abnormality that contraindicates regional anesthesia: INR >1.5, or platelet count <100,000/µL, or therapeutic anticoagulation that cannot be safely paused
* Infection at or near the needle insertion site
* Severe hepatic or renal impairment
* Chronic opioid therapy (>30 days of daily opioids before surgery)
* Cognitive impairment or delirium that prevents reliable pain assessment
* BMI >40 kg/m² (due to potential technical difficulty and reduced accuracy of ultrasound guidance)
* Previous regional block affecting the target area for the current surgery
* Pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia | Within 48 hours after surgery.
  Time (in hours) from completion of the PENG block to the first administration of a rescue analgesic (opioid or non-opioid) given for pain intensity ≥4 on the 0-10 Numerical Rating Scale (NRS).

SECONDARY OUTCOMES:
Pain Intensity at Rest (NRS 0-10) | 4 hours after surgery.
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups across predefined time points.
Pain Intensity at Rest (NRS 0-10) | 8 hours after surgery.
  ain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups across predefined time points.
Pain Intensity at Rest (NRS 0-10) | 12 hours after surgery.
  ain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups across predefined time points.
Pain Intensity at Rest (NRS 0-10) | 24 hours after surgery.
  ain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups across predefined time points.
Pain Intensity at Rest (NRS 0-10) | 48 hours after surgery.
  ain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups across predefined time points.
Pain Intensity During Movement (NRS 0-10) | 4 hours after surgery.
  Pain intensity during standardized hip movement (e.g., flexion or assisted mobilization) measured using the 0-10 Numerical Rating Scale.
Pain Intensity During Movement (NRS 0-10) | 8 hours after surgery.
  Pain intensity during standardized hip movement (e.g., flexion or assisted mobilization) measured using the 0-10 Numerical Rating Scale.
Pain Intensity During Movement (NRS 0-10) | 12 hours after surgery.
  Pain intensity during standardized hip movement (e.g., flexion or assisted mobilization) measured using the 0-10 Numerical Rating Scale.
Pain Intensity During Movement (NRS 0-10) | 24 hours after surgery.
  Pain intensity during standardized hip movement (e.g., flexion or assisted mobilization) measured using the 0-10 Numerical Rating Scale.
Pain Intensity During Movement (NRS 0-10) | 48 hours after surgery.
  Pain intensity during standardized hip movement (e.g., flexion or assisted mobilization) measured using the 0-10 Numerical Rating Scale.
Total Opioid Consumption | 0-24 hours and 0-48 hours after surgery.
  Cumulative dose of opioids converted to oral morphine milligram equivalents (MME).
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 4 hours after surgery.
  Quadriceps muscle strength will be assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the applied regional anesthesia techniques.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 8 hours after surgery.
  Quadriceps muscle strength will be assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the applied regional anesthesia techniques.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 12 hours after surgery.
  Quadriceps muscle strength will be assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the applied regional anesthesia techniques.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 24 hours after surgery.
  Quadriceps muscle strength will be assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the applied regional anesthesia techniques.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 48 hours after surgery.
  Quadriceps muscle strength will be assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the applied regional anesthesia techniques.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-48 hours after surgery.
  Presence of nausea or vomiting requiring antiemetic therapy. Proportion of patients with at least one episode will be recorded.
Hemodynamic Adverse Events | From block placement until 24 hours after surgery.
  Incidence of hypotension (systolic BP <90 mmHg or >30% decrease from baseline) and bradycardia (HR <50/min) requiring treatment.
Block-Related Adverse Events, Including Neurological Complications | From block placement until 30 days after surgery.
  Incidence of complications related to the PENG block or perineural adjuvants, including prolonged sensory or motor deficit, nerve injury (evaluated in outpatient clinic if required), hematoma, infection at the injection site, persistent weakness, or local anesthetic systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the results of this study will be made available to other researchers. Shared IPD will include demographic information, clinical outcomes, adverse events, and all primary and secondary outcome variables collected during the study. No information that could identify participants will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available beginning 12 months after publication of the primary results and will remain available for 5 years after publication.
Access Criteria: Data will be shared with qualified researchers for scientific purposes upon reasonable request. Requests will be evaluated by the study investigators. A data sharing agreement may be required.